CLINICAL TRIAL: NCT04088539
Title: Building Capacity and Promoting Smoking Cessation in the Correctional Institutions
Brief Title: Promoting Smoking Cessation in the Correctional Institutions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CSD 2019-2021
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Brief intervention; Correctional institution
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A (Experimental): CSD participants will receive a combined intervention:
  1. Brief intervention using AWARD advice at baseline,
  2. Video-based health education
  Interventions: Behavioral: AWARD advice; Behavioral: Video-based health education

INTERVENTIONS:
Behavioral: AWARD advice — Ask about smoking history, Warn about the high risk of smoking, Advise to quit as soon as possible, Refer to the smoking cessation services, and Do it again (if the smokers refused to set quit date)
Behavioral: Video-based health education — Educational videos on smoking and health will be developed to improve the knowledge of CSD smokers. The videos aim to raise their awareness on these important health topics and acquire effective cessation methods. The effectiveness of the educational videos will be evaluated by pre- and post-tests through a self-administered survey that assess the changes in knowledge related to smoking hazards, benefits of quitting, and methods to quit smoking.

SUMMARY:
The aim of this project is to promote and evaluate a smoking cessation intervention through the "Quit to Win" Contest organised in correctional institutions in Hong Kong.

The aim of this project is to promote and evaluate a smoking cessation intervention through the "Quit to Win" Contest organised in correctional institutions in Hong Kong. The specific objectives of the study are:

1. To test the effectiveness of face-to-face brief cessation advice and video education for smoking cessation among current smokers at the correctional institutions in Hong Kong;
2. To evaluate the process and outcome of the recruitment of smokers through qualitative interviews; and
3. To conduct qualitative interviews with quitters and non-quitters to examine their experience on the intervention.

DETAILED DESCRIPTION:
Although smoking prevalence is decreasing in Hong Kong, there are still 615,000 daily cigarette smokers in Hong Kong in 2017 and half will be killed by smoking [5] which accounts for over 7,000 deaths per year. Smoking is a highly addictive behavior and it is difficult for smokers with strong nicotine dependence to quit without assistance. Despite the low smoking rate in the general population, smoking prevalence remain high in the correctional institutions. Incarcerated prisoners suffer disproportionately from mental illness, substance use disorders and disease infections. They are in need of health care such as treatment or prevention for smoking. There is a lack of evidence on the effectiveness of smoking cessation intervention in the correctional setting. More work is required to provide smoking cessation assistance to these high risk and underserved population.

The aim of this project is to promote and evaluate a smoking cessation intervention through the "Quit to Win" Contest organised in correctional institutions in Hong Kong. The specific objectives of the study are:

1. To test the effectiveness of face-to-face brief cessation advice and video education for smoking cessation among current smokers at the correctional institutions in Hong Kong;
2. To evaluate the process and outcome of the recruitment of smokers through qualitative interviews; and
3. To conduct qualitative interviews with quitters and non-quitters to examine their experience on the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Smoke at least 1 cigarette per day in the past 3 months
* Able to communicate in Cantonese (including reading Chinese)
* Exhaled carbon monoxide (CO) 4 ppm or above, assessed by a validated CO smokerlyzer
* Intent to quit / reduce smoking

Exclusion Criteria:

* Smokers who have difficulties (either physical or cognitive condition) to communicate
* Currently following other smoking cessation programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical validated quit rate at 6-month follow-up | 6-month follow-up
  The primary outcome is biochemically validated quit rates (exhaled CO < 4 ppm and salivary cotinine < 10 ng/ml) at 6-month
Biochemical validated quit rate at 3-month follow-up | 3-month follow-up
  The primary outcome is biochemically validated quit rates (exhaled CO < 4 ppm and salivary cotinine < 10 ng/ml) at 3-month

SECONDARY OUTCOMES:
Smoking quit rate change from baseline at 3-month follow-up | 3-month follow-up
  Self-reported 7-day point prevalence (pp) quit rate at 3-month
Smoking quit rate change from baseline at 6-month follow-up | 6-month follow-up
  Self-reported 7-day point prevalence (pp) quit rate at 6-month
Smoking reduction rate change from baseline at 3-month follow-up | 3-month follow-up
  Rate of smoking reduction by at least half of baseline amount
Smoking reduction rate change from baseline at 6-month follow-up | 6-month follow-up
  Rate of smoking reduction by at least half of baseline amount

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided